CLINICAL TRIAL: NCT03597555
Title: A Randomized, Double-blind, Placebo-controlled Trial Comparing the Efficacy and Tolerance of Sodium Oxybate in Patients Affected With Idiopathic Hypersomnia
Brief Title: Sodium Oxybate in Idiopathic Hypersomnia
Acronym: SODHI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL17_0375
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Hypersomnia
Keywords: Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xyrem (Experimental): Xyrem (Sodium Oxybate), oral solution 500mg/mL First night after V1: Dose prescribed at 4.5 g per night (2.25 g x 2) for 2 weeks First night after V2: Dose increased to 6 g per night (3 g x 2) for 2 weeks, according to investigator's opinion, tolerance of drug and CGI-S First night after V3: Dose either maintained stable at 6 g or increased to 9 g per night (4.5 g x 2) with dose increments of 1.5 g per night (0.75 g x 2) every week, based on benefit-risk ratio, for 2 weeks.
  First night after V4: Dose maintained at 9 g or reduced at 6 g per night according to benefit-risk ratio for 2 weeks. No dose adjustment during the Maintenance period.
  First night after V5: Taper period. Dose decrease by 2.25 g x 2 every two days until complete withdrawal
  Interventions: Drug: Sodium Oxybate Oral Solution 500 MG/ML
- Placebos (Placebo Comparator): Xyrem Placebo: sodium citrate solution in equimolar concentration of sodium in the 500 mg/mL Xyrem oral solution, PH adjusted with malic acid
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Sodium Oxybate Oral Solution 500 MG/ML — First night after V1: Dose prescribed at 4.5 g per night (2.25 g x 2) for 2 weeks First night after V2: Dose increased to 6 g per night (3 g x 2) for 2 weeks, according to investigator's opinion, tolerance of drug and CGI-S First night after V3: Dose either maintained stable at 6 g or increased to 9 g per night (4.5 g x 2) with dose increments of 1.5 g per night (0.75 g x 2) every week, based on benefit-risk ratio, for 2 weeks.
  First night after V4: Dose maintained at 9 g or reduced at 6 g per night according to benefit-risk ratio for 2 weeks. No dose adjustment during the Maintenance period.
  First night after V5: Taper period. Dose decrease by 2.25 g x 2 every two days until complete withdrawal
  Arms: Xyrem
Drug: Placebos — Xyrem Placebo: sodium citrate solution in equimolar concentration of sodium in the 500 mg/mL Xyrem oral solution, PH adjusted with malic acid
  Arms: Placebos

SUMMARY:
this study evaluates of the efficacy of sodium oxybate on excessive daytime sleepiness using Epworth sleepiness scale over 8 weeks compared to placebo

DETAILED DESCRIPTION:
Bicentric, randomized, double-blind controlled study Outpatients aged from 18 to 60 years, suffering from current idiopathic hypersomnia (ICSD-3), recruited via medical consultations in the investigation centers Randomization in Xyrem or placebo arms after the inclusion visit,

1.Screening Period (up to 15 days), 2.Titration Period (up to 45 days), 3.Maintenance Period (minimum 15 days), 4.Safety Follow-Up Period (14 days)

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of idiopathic hypersomnia (ICSD-3 criteria)
* Age between 18 and 60 years-old
* BMI between 18 and 35 kg/m2
* MSLT: mean sleep latency (MSL) ≤8 minutes and < 2 SOREMPs, AND/OR total sleep time > 11h/24h on 24-hours long-term polysomnography
* Polysomnography recording: sleep efficiency > 85%, total sleep time ≥6 hours, AHI <10/hour, micro-arousals index <15/hour, PLM index associated with micro-arousals <10/hour.
* Absence of sleep deprivation, assessed by actigraphy or sleep logs
* ESS score ≥14 points
* Written informed consent
* National health insurance cover

Exclusion Criteria:

* Current alcohol intake or treatment with modafinil, amphetamine, methylphenidate, mazindol, pitolisant, neuroleptics, sedative hypnotics, barbiturates, general anesthetics, myorelaxants, other CNS depressants, antidepressants*, anxiolytic drugs, anticonvulsive therapy, topiramate, inhibitors of GHB dehydrogenase (i.e. valproate, ethosuximide, phenytoin), budipine, dopamine antagonist antiemetics (except domperidone), opioids, benzodiazepines, Z-drugs, MAO inhibitors, COMT inhibitors, or sedative antihistamines. If patient has received such therapy, a washout-period of at least 15 days, or equivalent to 5 half-lives of the drug, prior to the inclusion in the study is required before starting treatment in this study.

  *30 days for antidepressants
* Previous intake of sodium oxybate
* Succinic semialdehyde dehydrogenase deficiency, porphyria
* Other central nervous system diseases: neurodegenerative diseases, seizure disorders or history of head trauma associated with loss of consciousness
* Lifetime history of suicide attempt or suicidal ideation in the past 6 months, prior history of psychotic episodes, current or recent history of a major depressive disorder (DSM-V), Beck depression inventory (BDI) > 16 and/or item G> 0
* History of chronic alcohol or drug abuse within the prior 12 months
* Malignant neoplastic disease requiring therapy within 12 months prior to Visit 1 or clinically relevant
* Heart failure, severe hypertension or other cardiovascular disease compromising the patient's wellbeing or ability to participate in this study
* Renal or hepatic impairment Compromised respiratory function
* Sleep-related breathing disorders (AHI ≥ 10/h)
* No regular sleep at night: shift work or other continuous non-disease-related life conditions
* Participation in another study of an investigational drug within the 28 days prior to Visit 1 or currently
* Hypersensitivity to any of the components of the study medication
* Pregnancy (βHCG positive) and breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) score at the end-point visit | over 8 weeks
  Evaluation of difference in sleepiness with ESS between the 2 groups. ESS scores range from 0 to 24; there is a risk of pathological daytime sleepiness if score is > 10.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dauvilliers Y, Chenini S, Thobois O, Rassu AL, Denis C, Guiraud L, Jaussent I, Barateau L. Efficacy and Safety of Sodium Oxybate in Adults With Idiopathic Hypersomnia: A Randomized Controlled Trial. Neurology. 2025 Jun 10;104(11):e213690. doi: 10.1212/WNL.0000000000213690. Epub 2025 May 13. PMID 40359459